CLINICAL TRIAL: NCT03143452
Title: Comparison Between 2% Lidocaine Gel and 5% Tetracaine Eye Drop as Topical Anesthesia in Phacoemulsification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Susilo Chandra, Anesthesiologist Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes015
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Adult Patients Undergoing Phacoemulsification With Topical Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine gel (Active Comparator): Lidocaine gel group: received 2% lidocaine gel in 1 ml syringe, applied to the eye 5 minutes before phacoemulsification
  Interventions: Drug: lidocaine gel
- tetracaine eye drop (Active Comparator): Tetracaine eye drop group: received 0.5% tetracaine eye drop 5 minutes before phacoemulsification
  Interventions: Drug: tetracaine eye drop

INTERVENTIONS:
Drug: lidocaine gel — 2% lidocaine gel in 1 ml syringe, applied to the eye 5 minutes before phacoemulsification
  Arms: lidocaine gel
Drug: tetracaine eye drop — 0.5% tetracaine eye drop was given 5 minutes before phacoemulsification
  Arms: tetracaine eye drop

SUMMARY:
This study aimed to compare the efficacy between 2% lidocaine gel vs 0.5% tetracaine eye drop as topical anesthesia in phacoemulsification

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study and randomized into two groups (Lidocaine gel and tetracaine eye drop group). Lidocaine group received 2% lidocaine gel in 1 ml syringe, applied to the eye. Tetracaine group received 0.5% tetracaine eye drop. Topical anesthesia was given 5 minutes before phacoemulsification. Five minutes after phacoemulsification finished, visual analog score (VAS) and subjects and surgeon's satisfaction were assessed. Every additional topical anesthesia needed was recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients aged more than 40 years old who were planned to undergo elective phacoemulsification with intraocular lens implantation at operating room. The surgery was operated by an experienced ophthalmologist. Subjects had been explained about the study, and agreed to enroll and have signed the informed consent form.

Exclusion Criteria:

* Subjects with history of allergy to topical anesthesia (2% lidocaine gel and 0.5% tetracaine eye drop), subjects who used another method of intraoperative anesthesia other than topical anesthesia, subjects with history of phacoemulsification before, subjects with difficulty in communication, dementia, and anxiety.

Dropout Criteria:

* Phacoemulsifications duration more than 30 minutes, and subjects who resigned from the study before the study ended

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | Day 1
  assessing subject's pain with visual analog scale

SECONDARY OUTCOMES:
Additional topical anesthesia requirement | Day 1
  Number of additional topical anesthesia given after the first dose
Subjects and surgeon's satisfactory | Day 1
  Assessment is done using questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jinapriya D, Almeida DR, Johnson D, Irrcher I, El-Defrawy SR. Anaesthetic plus dilating gel improves pupil dilation for cataract surgery. Can J Ophthalmol. 2012 Apr;47(2):145-9. doi: 10.1016/j.jcjo.2012.01.007. Epub 2012 Mar 14. PMID 22560419
- [Background] Tsoumani AT, Asproudis IC, Damigos D. Tetracaine 0.5% eyedrops with or without lidocaine 2% gel in topical anesthesia for cataract surgery. Clin Ophthalmol. 2010 Sep 7;4:967-70. doi: 10.2147/opth.s11755. PMID 20856590
- [Background] Waheeb S. Topical anesthesia in phacoemulsification. Oman J Ophthalmol. 2010 Sep;3(3):136-9. doi: 10.4103/0974-620X.71892. PMID 21120050
- [Background] Chalam KV, Murthy RK, Agarwal S, Gupta SK, Grover S. Comparative efficacy of topical tetraVisc versus lidocaine gel in cataract surgery. BMC Ophthalmol. 2009 Aug 17;9:7. doi: 10.1186/1471-2415-9-7. PMID 19686592
- [Background] Shiroma HF, Shimono KE, Farah ME, Goldhardt R, Grumann A Jr, Rodrigues EB. Comparative Study Between Lidocaine Gel 2% and 5% for Ophthalmic Procedures. J Ocul Pharmacol Ther. 2016 May;32(4):192-5. doi: 10.1089/jop.2015.0002. Epub 2016 Jan 20. PMID 26790036
- [Background] Rafailov L, Kulak A, Weedon J, Shinder R. Comparison of Lidocaine Gel-Assisted Transconjunctival and Transcutaneous Local Anesthesia for Outpatient Eyelid Surgery. Ophthalmic Plast Reconstr Surg. 2015 Nov-Dec;31(6):470-3. doi: 10.1097/IOP.0000000000000391. PMID 25675169
- [Background] Soliman MM, Macky TA, Samir MK. Comparative clinical trial of topical anesthetic agents in cataract surgery: lidocaine 2% gel, bupivacaine 0.5% drops, and benoxinate 0.4% drops. J Cataract Refract Surg. 2004 Aug;30(8):1716-20. doi: 10.1016/j.jcrs.2003.12.034. PMID 15313296
- [Background] Shah H, Reichel E, Busbee B. A novel lidocaine hydrochloride ophthalmic gel for topical ocular anesthesia. Local Reg Anesth. 2010;3:57-63. doi: 10.2147/lra.s6453. Epub 2010 Aug 10. PMID 22915870
- [Background] Amiel H, Koch PS. Tetracaine hydrochloride 0.5% versus lidocaine 2% jelly as a topical anesthetic agent in cataract surgery: comparative clinical trial. J Cataract Refract Surg. 2007 Jan;33(1):98-100. doi: 10.1016/j.jcrs.2006.09.013. PMID 17189801
- [Background] Irle S, Luckefahr MH, Tho Seeth T. [Tetracaine drops versus lidocaine gel for topical anaesthesia in cataract surgery]. Klin Monbl Augenheilkd. 2003 Sep;220(9):625-8. doi: 10.1055/s-2003-42811. German. PMID 14533061